CLINICAL TRIAL: NCT06184698
Title: Liposomal Irinotecan + Leucovorin + 5-fluorouracil + Bevacizumab as Second-line Therapy in Metastatic Colorectal Cancer (IRIS)：a Multicenter, Single-arm, Prospective, Phase II Study
Brief Title: Liposomal Irinotecan and Leucovorin/5-fluorouracil Plus Bevacizumab in Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K04
Record Dates: First submitted 2023-12-12; First posted 2023-12-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: liposomal irinotecan; second-line therapy; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): liposomal irinotecan+5-FU/LV+ bevacizumab q2w
  Interventions: Drug: liposomal irinotecan; Drug: 5-FU; Drug: LV; Drug: Bevacizumab

INTERVENTIONS:
Drug: liposomal irinotecan — liposomal irinotecan 70 mg/m²
  Other Names: nal-IRI
Drug: 5-FU — 5-FU 2400 mg/m²
  Other Names: Fluorouracil
Drug: LV — 5-FU 2400 mg/m²
  Other Names: Calcium folinate
Drug: Bevacizumab — bevacizumab 5 mg/kg
  Other Names: Avastin

SUMMARY:
This is a multi-center, single-arm study to investigate the efficacy and safety of liposomal irinotecan+5-FU/LV+ bevacizumab as second-line therapy in metastatic colorectal cancer in Chinese population.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) has a poor prognosis and poses a serious threat to human health. FOLFIRI (irinotecan+5-FU/LV) / FOLFOX (oxaliplatin+5-FU/LV) ± angiogenesis inhibitors are common treatments for advanced CRC. For patients receiving oxaliplatin-based therapy, irinotecan-based therapy is recommended as second-line therapy. Liposomal irinotecan is a new pharmaceutical form of traditional irinotecan. It adopts a special loading technology to encapsulate traditional irinotecan in liposomes, which can avoid its hydrolysis under physiological conditions, increase the affinity with cancer cells, overcome drug resistance, increase the drug uptake by cancer cells, reduce the drug dose, improve the efficacy and reduce the toxic side effects. The aim of this study is to explore the efficacy and safety of liposomal irinotecan+5-FU/LV + bevacizumab as second-line treatment for metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old.
* Histologically or cytologically proven colon or rectum adenocarcinoma.
* Confirmed as unresectable metastatic disease through radiological examination.
* At least one measurable lesion (according to RECIST v1.1).
* First-line treatment with oxaliplatin-based therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 2.
* The expected survival time ≥3 months.
* Subject has adequate biological parameters as demonstrated by the following: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin (Hgb) ≥90 g/L, white blood cell (WBC)≥3.0×10^9/L.
* Adequate hepatic function as evidenced by total bilirubin ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and alanine aminotransferase (ALT) ≤2.5 x ULN, ≤5 x ULN if liver metastases are present.
* Adequate renal function as evidenced by serum creatinine (Cr)≤1.5 x ULN or creatinine clearance ≥60 mL/min, proteinuria <2+.
* Normal coagulation function (INR≤1.5).
* Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening.

Exclusion Criteria:

* Any other malignancy within 5 years prior to randomization, with the exception of cured in-situ carcinoma or basal cell carcinoma.
* Previous treatment with irinotecan/liposomal irinotecan.
* MSI-H/dMMR
* Massive pleural effusion or ascites requiring intervention.
* Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
* Active HIV, HBV, HCV infection.
* Combined with uncontrollable systemic diseases.
* Presence of severe gastrointestinal disease (including active bleeding, > grade 1 obstruction , > grade 1 diarrhea or gastrointestinal perforation)
* History of laparotomy, thoracotomy, or intestinal resection within 28 days before enrolment.
* Presence of interstitial pneumonia or pulmonary fibrosis.
* Allergy to or intolerance to therapeutic drugs or their excipients;.
* History of pulmonary hemorrhage/hemoptysis ≥ Grade 2 (defined as bright red blood of at least 2.5mL) within one month prior to enrollment.
* Presence of arterial embolism, severe bleeding (excluding bleeding caused by surgery) or tendency for existing embolism or severe bleeding within 6 months before enrollment.
* Patients with symptomatic central nervous system metastases.
* Documented serum albumin ≤3 g/dL
* Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1.
* Pregnant or breastfeeding women, or subjects of childbearing age who refuse contraception.
* Participated in other trial within 30 days prior to the first dose of study treatment.
* Patients who had received any intravenous antineoplastic therapy within 28 days or oral antineoplastic therapy within 14 days before the first dose of study drug
* Patients who are not suitable to participate in this trial for any reason judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate | 4 months
  Defined as the percentage of patients who achieved CR, PR, and stable disease (SD) according to RECIST v1.1.
Duration of Response | 4 months
  Defined as the time from the initiation of a response (first confirmation of CR or PR) to disease progression or death from any cause, whichever occurred first.
Progress-free survival | 6 months
  Defined as time from the subject's enrollment to first documented disease progression using RECIST version 1.1 by investigator review or death due to any cause, whichever occurred first.
Overall survival | 1 year
  Defined as the time between signing the informed consent form and death due to various causes.
Incidence of adverse events | 5 months
  Use NCI-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Overall Officials: Guiying Wang, Professor, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No